CLINICAL TRIAL: NCT04710550
Title: Exploring the Utility of [18F]3F4AP for Demyelination Imaging in Controls, Neurodegeneration and Traumatic Brian Injury
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Marc D.Normandin, Ph.D, Associate Professor, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020P002254
Record Dates: First submitted 2020-12-17; First posted 2021-01-14 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Brain Injuries, Traumatic; Demyelinating Disorder; Alzheimer Disease
Keywords: 3F4AP
MeSH Terms: conditions — Brain Injuries, Traumatic; Demyelinating Diseases; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Safety/Dosimetry Cohort (Experimental)
  Interventions: Drug: F18-3F4AP
- Traumatic Brain Injury (Experimental)
  Interventions: Drug: F18-3F4AP
- AD/MCI (Experimental)
  Interventions: Drug: F18-3F4AP
- Healthy Controls (Active Comparator)
  Interventions: Drug: F18-3F4AP

INTERVENTIONS:
Drug: F18-3F4AP — PET Scan

SUMMARY:
The overall objective is to obtain an initial assessment of the value of using [18F]3F4AP for imaging demyelinating diseases such as traumatic brain injury (TBI), neurodegenerative diseases such as mild cognitive impairment (MCI) and Alzheimer's Disease (AD):

* Aim 1) Assess the safety of [18F]3F4AP in healthy volunteers and subjects with traumatic brain injury (TBI) and neurocognitive impaired subjects (AD/MCI). Hypothesis 1: Administration of [18F]3F4AP will result in no changes in vitals or other adverse events.
* Aim 2) Assess the radiation doses to the main organs in healthy volunteers. Hypothesis 2: the radiation doses to each organ will be comparable in all subjects and within the acceptable limits.
* Aim 3) Assess the pharmacokinetics of a bolus infusion of [18F]3F4AP in humans including healthy volunteers and patients. Hypothesis 3: the pharmacokinetics of [18F]3F4AP at the whole brain level will be similar in controls, TBI and AD/MCI subjects. The kinetics in demyelinated lesions will be slower than in healthy areas.
* Aim 4) Correlate MR images with [18F]3F4AP PET images. Hypothesis 4A: all the lesions seen on the MRI will show increased signal (VT or SUV) on the PET images. Hypothesis 4B: some of the lesions on the MRI will show increased signal (VT or SUV) on the PET but not all.
* Aim 5) Correlate [18F]3F4AP PET signal with neuropsychological testing in people with TBI and AD/MCI. Hypothesis 5A: increased PET signal (VT or SUV) will correlate with impaired Mini Mental State Examination (MMSE).

ELIGIBILITY:
Inclusion Criteria:

* Subjects are 18 years of age and older, except AD subjects who are 60 to 90 years of age.

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the exclusion criteria for PET/CT or MRI studies applies. A negative STAT quantitative serum hCG pregnancy test is required on the day of the PET/CT scan before female subjects of childbearing potential can participate. Any woman of childbearing potential, who is seeking to become pregnant, is breastfeeding, or who suspects she may be pregnant will not be enrolled in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 5 years
  Determine number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Marc Normandin, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramos-Torres K, Sun Y, Takahashi K, Zhou YP, Brugarolas P. Common anesthetic used in preclinical PET imaging inhibits metabolism of the PET tracer [18F]3F4AP. J Neurochem. 2024 Sep;168(9):2577-2586. doi: 10.1111/jnc.16118. Epub 2024 May 1. PMID 38690718